CLINICAL TRIAL: NCT04908358
Title: The Wandering Nerve: Gateway to Boost Alzheimer's Disease Related Cognitive
Brief Title: The Wandering Nerve: Gateway to Boost Alzheimer's Disease Related Cognitive Performance
Acronym: WALLe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Heidi Jacobs, Associate Professor of Radiology, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2021P000498; 1R01AG068062-01A1 (NIH)
Record Dates: First submitted 2021-05-04; First posted 2021-06-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Aging
Keywords: Transcutaneous vagus nerve stimulation; Memory; Brainstem; Aging; Preclinical Alzheimer's disease

STUDY DESIGN:
Intervention Model Description: Randomized cross-over followed by placebo-controlled study (allocation to placebo or control condition takes APOE-E4 status into account and the previous ordering of the cross-over design)
Who Masked: Participant
Masking Description: Participant will not be informed of condition. The investigators will work with blinded data (but can know the condition during intervention)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sham preceded by cross-over Sham-Stimulation (Sham Comparator): Cross-over: Sham followed by experimental Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) Wash-out period of four weeks Ten daily sessions of sham during 2 weeks
  Interventions: Other: Sham transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions
- Sham preceded by cross-over Stimulation-Sham (Sham Comparator): Cross-over: experimental Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) followed by Sham Wash-out period of four weeks Ten daily sessions of sham during 2 weeks
  Interventions: Other: Sham transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions
- Stimulation preceded by cross-over Sham-Stimulation (Experimental): Cross-over: Sham followed by experimental Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) Wash-out period of four weeks Ten daily sessions of RAVANS during 2 weeks
  Interventions: Other: Active transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions
- Stimulation preceded by cross-over Stimulation-Sham (Experimental): Cross-over: experimental Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) followed by sham Wash-out period of four weeks Ten daily sessions of RAVANS during 2 weeks
  Interventions: Other: Active transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions
- cross-over Stimulation-Sham (Other): Cross-over: experimental Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) followed by sham One time RAVANS versus one time Sham Two weeks wash-out
  Interventions: Other: Active transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions; Other: Sham transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions
- cross-over Sham-Stimulation (Other): Cross-over: Sham followed by experimental Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) One time RAVANS versus one time Sham Two weeks wash-out
  Interventions: Other: Active transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions; Other: Sham transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions

INTERVENTIONS:
Other: Active transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions — Stimulation of vagus nerve in the outer ear
  Other Names: Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS); transcutaneous vagus nerve stimulation
  Arms: Stimulation preceded by cross-over Sham-Stimulation; Stimulation preceded by cross-over Stimulation-Sham; cross-over Sham-Stimulation; cross-over Stimulation-Sham
Other: Sham transcutaneous vagus nerve stimulation respiratory-gated non-painful electrical stimulation of the auricle for 10 minute sessions — Sham stimulation of vagus nerve in the outer ear
  Other Names: Sham Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS); Sham transcutaneous vagus nerve stimulation
  Arms: Sham preceded by cross-over Sham-Stimulation; Sham preceded by cross-over Stimulation-Sham; cross-over Sham-Stimulation; cross-over Stimulation-Sham

SUMMARY:
In this research study the investigators want to find out if a non-invasive electrical brain stimulation method called RAVANS (also called tVNS) can have a beneficial effect on cognition in older individuals. The investigators also want to understand whether certain individual factors contribute to the effect of RAVANS on cognition. RAVANS is only used in research studies.

DETAILED DESCRIPTION:
The intervention will be studied in 140 older individuals using a randomized cross-over design of sham versus RAVANS stimulation (2 sessions separated by 4 weeks) during a functional magnetic resonance imaging (fMRI) task. Participants will then be randomized to daily tVNS or sham sessions during 10 visits within two weeks, and two follow-up cognitive assessments each after 2 months of the last intervention session. The face-name association task will be the main outcome measure. The investigators will also draw blood twice to examine whether the response on the outcome is dependent on Alzheimer's disease related biomarker, and whether RAVANS has effects on inflammatory responses.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Willingness and ability to comply with scheduled visits, magnetic resonance imaging (MRI) scanning, laboratory tests, and other study procedures.
* Subjects with well-controlled vascular risk factors, such as treated hypertension, treated hyperlipidemia or well controlled Type II diabetes will be included.
* Stable medications for at least 30 days.
* Mini Mental State Exam adjusted for age and education of 25 to 30, inclusive or a Telephone Interview for Cognitive Status score of at least 32
* Perform within 1.5 S.D. of age and education matched norms on the Logical Memory Paragraph Delayed Recall
* Geriatric Depression Scale < 11
* Aged 60-85, inclusive
* Right-handed
* Reduced vision is allowed if it can be corrected with MRI-goggles

Exclusion Criteria:

* Prior known diagnosis of mild cognitive impairment (MCI) or dementia
* Use of investigational drugs or devices within 60 days prior to screening
* Subjects with contraindications to MRI cannot participate (i.e., implanted metal including pacemakers, cerebral spinal fluid shunts, aneurysm clips, artificial heart valves, ear implants or metal/foreign objects in the eyes and those with a history of claustrophobia)
* Pregnant.
* Major psychiatric disorders such as schizophrenia, schizoaffective disorder, major affective disorder in mid-life, or treatment with electroconvulsive therapy (ECT) (Mild depression that is well treated with stable dose of selective serotonergic reuptake inhibitor (SSRI) antidepressants will be allowed).
* Have a history of major head trauma defined as a loss of consciousness and/or trauma requiring hospitalization
* Substance abuse within the past 2 years
* Active hematological, renal, pulmonary, endocrine or hepatic disorders.
* Evidence of cortical infarcts or strategically placed lacunar infarct (e.g. dorsal medial nucleus of thalamus). MRI evidence of mild white matter signal abnormalities will be allowed.
* Active cancer, metabolic encephalopathy, infection
* Active cardiovascular disease, stroke, congestive or severe heart failure
* Huntington's disease, hydrocephalus or seizure disorder
* Cataracts, glaucoma, detached retina's, eye surgery involving the muscles; droopy eyelids, penetrating eye wounds and use of anticholinergic eye drop use
* Weight equal to or greater than 300 lbs (weight limit of the MRI table).
* Recurrent vaso-vagal syncopal episodes
* Unilateral or bilateral vagotomy
* Severe valvular disorder (i.e. prosthetic valve or hemodynamically relevant valvular diseases)
* Sick sinus syndrome
* Hypotension due to autonomic dysfunction

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Performance on the Face-name association memory task (FNAME) | Up to 25 weeks: assessed during week 1, week 2, week 8,week 9, week 17 and week 25
  Change from baseline at each visit where FNAME is completed: Scores are z-scores with a mean of zero. Higher scores are better (there is no minimum/maximum).
Being a responder as determined by Face-name association memory task (FNAME) change scores | Based on data from the first 4 weeks (cross-over)
  Participants are grouped in being a responder (1) or non-responder (0).

SECONDARY OUTCOMES:
Performance on other cognitive composite scores: this includes a composite score of memory, a composite score of executive function and the Preclinical Alzheimer's disease cognitive composite. | Up to 25 weeks: assessed during week 1, week 2, week 8,week 9, week 17 and week 25
  Change from baseline at each visit where neuropsychological data is collected. Composites are calculated following a confirmatory factor analyses. All scores (correct answers) will be expressed in z-scores and higher scores are better (there is no minimum/maximum).
Change in inflammatory responses (aggregated) | Assessed during the first week and during week 9
  Change from baseline to after intervention, these markers will be analyzed from blood:
  * Interleukins (IL): IL-1β, IL-2, IL-6, IL-8
  * Tumor necreose factor alpha (TNF-α)
  * Macrophage inflammatory protein (MIP1B)
  * Monocyte chemoattractant protein (MCP-1)
  * Complement components: C1q and C3
  * soluble triggering receptor expressed on myeloid cells (TREM2).
  Following stability analyses, specific markers will be selected (with advise by Dr. Arnold) and analysed individually (see outcome measures 5-10) and in aggregated form (here). Markers will be combined following a principal component analyses and will be normalised. Values will be expressed in z-scores.
Change in inflammatory responses (interleukins) | Assessed during the first week and during week 9
  Change from baseline to after intervention:
  - Interleukins (IL): IL-1β, IL-2, IL-6, IL-8 (expressed in IU, international units)
Change in inflammatory responses (TNF) | Assessed during the first week and during week 9
  Change from baseline to after intervention:
  - Tumor necreose factor alpha (TNF-α) (units/ml)
Change in inflammatory responses (MIP) | Assessed during the first week and during week 9
  Change from baseline to after intervention:
  - Macrophage inflammatory protein (MIP1B) (units/ml)
Change in inflammatory responses (MCP) | Assessed during the first week and during week 9
  Change from baseline to after intervention:
  -Monocyte chemoattractant protein (MCP-1) (units/ml)
Change in inflammatory responses (C) | Assessed during the first week and during week 9
  Change from baseline to after intervention:
  - Complement components: C1q and C3 (units/ml)
Change in inflammatory responses (TREM) | Assessed during the first week and during week 9
  Change from baseline to after intervention:
  - soluble triggering receptor expressed on myeloid cells (sTREM2) (units/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi IL Jacobs, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with NIH regulations, as provided in the manual of the NIH (SF424 (R&R)), data will be made available at the time of publication of the primary results or within 9 months of database lock, whichever comes first. A more detailed plan for sharing data and a data user agreement procedure will be set up during the study.
Supporting Information: Study Protocol, ICF
Time Frame: Consistent with NIH regulations, as provided in the manual of the NIH (SF424 (R&R)), data will be made available at the time of publication of the primary results or within 9 months of database lock, whichever comes first, and will be available for at least 3 years or until the sharing platform is no longer available. A more detailed plan for sharing data and a data user agreement procedure will be set up during the study.
Access Criteria: Access to the clinical trial IPD can be requested by qualified scientists affiliated a research institutions, and will be provided following review and approval of a research proposal, statistical analysis plan and after signing a data user agreement. Requests can be submitted to wallestudy@mgh.harvard.edu from the first publication date of the primary results or within 9 months of database lock, whichever comes first. In the future, more information on data requests can be found on http://www.heidijacobs.org/. A more detailed plan for sharing data and a data user agreement procedure will be set up during the study.
URL: http://www.heidijacobs.org